CLINICAL TRIAL: NCT00859235
Title: Predicting Oral Care Before Percutaneous Endoscopic Gastrostomy (PEG). The Influence of Oral Hygiene on Local Wound and Systemic Infection in Patients With PEG Placement
Brief Title: The Influence of Oral Hygiene on Local Wound and Systemic Infection in Patients With Percutaneous Endoscopic Gastrostomy Placement
Acronym: PEG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Zvi Fireman MD /head, Gasstroenterology Dept., Hillel Yaffe Med. Ctr.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HY022009
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Dysphagia; Peristomal Wound Infection
Keywords: Percutaneous endoscopic gastrostomy; peristomal wound infection; antibiotic mouth wash solution; prophylaxis prior Percutaneous endoscopic gastrostomy (PEG)
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Chlorhexidine gluconate 0.2%
- 2. Plain water (Placebo Comparator)
  Interventions: Other: Plain water

INTERVENTIONS:
Drug: Chlorhexidine gluconate 0.2% — Mouth wash prior to procedure
  Arms: 1
Other: Plain water — Mouth wash prior to procedure
  Arms: 2. Plain water

SUMMARY:
Percutaneous endoscopic gastrostomy (PEG) is commonly used for long term enteral feeding of patients with severe dysphagia. The most common complication is peristomal wound infection. The possible mechanism the bacterial from the oral cavity disseminate during the PEG insertion through the stomach to the abdominal wall, in spite the routine use of antibiotic prophylaxis, have reported low rates of wound infection in patients who were already receiving antibiotics at the time of PEG Our hypothesis that washing the oral cavity with antibiotic solution prior the insertion PEG , We planned a prospective, randomised, double blind, one centre study of antibiotic mouth wash solution (0.2% Chlorhexidine gluconate) as.prophylaxis in PEG

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo PEG

Exclusion Criteria:

* Previous GI surgery
* Coagulopathy
* Sepsis

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Assess impact mouth wash (containing 0.2% Chlorhexidine gluconate) (Taro Pharmaceutical Industries Haifa Israel) prior PEG insertion. | One month

SECONDARY OUTCOMES:
Follow the peristomal wound infection in patients who had prepared by mouth wash to a group a patients without mouth washing. | One month